CLINICAL TRIAL: NCT01939379
Title: Adductor Canal Nerve Block Following Total Knee Arthroplasty: A Randomized, Prospective Study Comparing High vs. Low Volume Bolus of 0.33% Ropivacaine
Brief Title: Adductor Canal Nerve Block Following Total Knee Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution. Efforts made to contact PI unsuccessful. No study data available.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 5130183
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Post-op Pain
Keywords: Total knee arthroplasty; nerve block; Pain control after surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 15ml ropivacaine (Active Comparator): Depending on what dose of ropivacaine the subject is randomized to he/she could receive the 15ml dose injected into the catheter every 6 hours
  Interventions: Drug: Morphine PCA started at the end of surgery, 1 Percocet 1/325mg every 4 hours; may receive a second Percocet if needed.
- 30ml ropivacaine (Active Comparator): If the subject is randomized to 30ml ropivacaine he/she will be injected through the catheter every 6 hours.
  Interventions: Drug: For the 30ml ropivacaine the intervention would be the subject can request extra pain medication which would be Percocet and/or morphine PCA.

INTERVENTIONS:
Drug: Morphine PCA started at the end of surgery, 1 Percocet 1/325mg every 4 hours; may receive a second Percocet if needed.
  Arms: 15ml ropivacaine
Drug: For the 30ml ropivacaine the intervention would be the subject can request extra pain medication which would be Percocet and/or morphine PCA.
  Arms: 30ml ropivacaine

SUMMARY:
The purpose of this study is that an adductor canal nerve block (putting numbing medicine near the nerve) has been shown to produce excellent pain relief with less pain medication use after knee replacement surgery.The investigators will be comparing the amount of pain relief following knee replacement surgery when you have a nerve block in place. There will be approximately 66 subjects participating in this study. After surgery subjects will receive numbing medication every 6 hours for 48 hours. Subjects will also receive a morphine PCA (patient controlled analgesia) after surgery and pain medication by mouth every 4 hours around the clock with the option to receive more pain medication if needed. Subjects will participate in the study up to 3 days.

ELIGIBILITY:
Inclusion Criteria:

1. Is the subject undergoing primary unilateral total knee arthroplasty?
2. Is the subject 18 to 99 years of age?
3. Is the subject ASA class 1, 2, or 3?
4. Does the subject have a BMI less than 35?
5. Can the subject consent in the English language?

Exclusion Criteria:

1. Does subject have an allergy to drugs used in this study;
2. Does subject have a daily intake of opiate medications that are considered stronger than hydrocodone?
3. Does subject have a history of alcohol or drug abuse
4. Has subject had a previous total knee arthroplasty?
5. Has subject had any neurologic deficits in the lower extremity being studied?

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Total Opiate pain medication | The total amount of opiate pain medication will be recorded at 6 hour intervals for 48 hours after surgery.
  At the end of the 48 hours period the total opiate pain medication taken will be collected and used for comparison as our primary outcome

SECONDARY OUTCOMES:
Patient satisfaction with pain control | We will look at the secondary outcome measure beginning every six hours for 48 hours after surgery
  Secondary outcome measures will include demographic characteristics, pain scores, medication administration,patient satisfaction with pain control and any complications that may have arisen. We will also record the location of the adductor canal catheter on the final bolus dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Medical Center East Campus Hospital, Loma Linda, California, United States